CLINICAL TRIAL: NCT06705309
Title: The Effect of a Web-Based Education Program and Educational Booklet Developed on Cervıcal Cancer on Women's Prevention Methods
Brief Title: Web-Based Education Program and Educational Booklet Developed on Cervıcal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Şen, Phd Student - Lecturer, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Istanbul UniversityC
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer Awareness, Prevention, HPV, Pap Smear
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-Based Education Group (Experimental): Web-Based Education Group
  Interventions: Behavioral: Web-Based Education

INTERVENTIONS:
Behavioral: Web-Based Education — The Effect of a Web-Based Education Program and Educational Booklet Developed on Cervıcal Cancer on Women's Prevention Methods

SUMMARY:
Cervical cancer is the fourth most common cancer type among women worldwide and ranks ninth in Turkey, making it the second most common gynecological cancer. The prevention of cancer heavily relies on identifying risk factors, implementing preventive measures, and early diagnosis. Cervical cancer is associated with high-risk Human Papilloma Virus (HPV) infections, transmitted primarily through sexual contact, accounting for 99.7% of cases. Risk-enhancing factors include early sexual activity, poor hygiene, low socioeconomic status, and immunosuppressive conditions. The World Health Organization (WHO) launched the "Cervical Cancer Elimination Program" to address this public health issue, aiming for 90% of girls to be vaccinated against HPV by age 15, 70% of women aged 35-45 to be screened, and 90% of women diagnosed with cancer to have access to treatment by 2030. The low participation rate in cervical cancer screening programs in Turkey highlights the urgent need to increase public awareness. Web-based education is an effective tool for promoting health behaviors and increasing awareness. Its cost-effectiveness, ability to reach large audiences, and easy accessibility make it a valuable resource in healthcare. Studies in the literature demonstrate that web-based and video-based education significantly enhance cervical cancer awareness and encourage pap smear test uptake. This study developed a web-based education program and an educational booklet on cervical cancer, based on the Health Belief Model, to evaluate their impact on women's knowledge, attitudes, and behaviors. The study aims to contribute to the dissemination of cervical cancer prevention methods and enrich the existing literature.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer among women worldwide and ranks ninth in Turkey, making it the second most common gynecological cancer. This highlights the significance of cervical cancer both globally and within Turkey. The prevention of this cancer is heavily reliant on identifying risk factors, implementing effective preventive measures, and ensuring early diagnosis. These factors play a crucial role in reducing the incidence of cervical cancer and improving the outcomes for affected individuals.

Cervical cancer is primarily associated with high-risk Human Papilloma Virus (HPV) infections, which are transmitted mainly through sexual contact. In fact, 99.7% of cervical cancer cases are linked to HPV infection. Understanding the risk factors for HPV and cervical cancer is essential for prevention. These risk-enhancing factors include early sexual activity, poor hygiene practices, low socioeconomic status, and immunosuppressive conditions, such as HIV infection or the use of immunosuppressive drugs.

To tackle this significant public health issue, the World Health Organization (WHO) launched the "Cervical Cancer Elimination Program," which sets ambitious goals to reduce the burden of cervical cancer by 2030. These goals include 90% of girls vaccinated against HPV by age 15, 70% of women aged 35-45 screened for cervical cancer, and 90% of women diagnosed with cervical cancer to have access to treatment. These targets are part of a broader effort to eliminate cervical cancer as a public health problem, aiming for a world where the incidence of cervical cancer is significantly reduced through vaccination, screening, and treatment accessibility.

Despite global efforts, there is a low participation rate in cervical cancer screening programs in Turkey, highlighting the urgent need to increase public awareness about the importance of early detection. Increasing awareness through educational campaigns can improve participation and, in turn, help reduce the incidence of cervical cancer.

Web-based education is increasingly recognized as an effective tool for promoting health behaviors and raising awareness on various health topics. Its key advantages include cost-effectiveness, accessibility, and convenience. Web-based programs are generally more affordable than in-person interventions and can reach a wide audience, including individuals who may not have easy access to healthcare facilities. Participants can engage with the content at their own pace, making it an attractive option for health education.

Studies have shown that web-based and video-based education can significantly enhance awareness about cervical cancer and encourage women to undergo preventive screenings, such as the Pap smear test, which is crucial for early detection.

The study developed a web-based education program and an educational booklet on cervical cancer, grounded in the Health Belief Model. This model focuses on individuals' perceptions of health risks and the benefits of taking preventive actions. The study aims to evaluate the impact of these educational tools on women's knowledge, attitudes, and behaviors regarding cervical cancer prevention. By assessing the effectiveness of these educational resources, the study aims to contribute to the dissemination of cervical cancer prevention methods and enrich the existing literature on the topic.

This research aims to provide valuable insights into how web-based education and educational booklets can be used to improve women's understanding of cervical cancer and enhance preventive behaviors. By contributing to public awareness and facilitating access to information, this study supports global and national efforts to reduce the burden of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30-65,
* Having never had a cervical cancer screening before,
* Having received training on cervical cancer,
* There is no obstacle to answering the questions physically, mathematically or spiritually,
* Having internet access,
* Being able to use a computer and/or tablet effectively,
* Academicians working in health programs,
* Healthy female academics who did not agree to participate in the research,
* Being able to use a computer

Exclusion Criteria:

* The emergence of any health problem that prevents the person from continuing the research,
* Not completing any of the required forms,
* Those who give up participating in the study at any stage of the study
* Do not visit 80% of the tabs in the web training program,
* Those who have never read the training booklet will be excluded.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Informing and Protecting Women About Cervical Cancer
Enrollment: 128 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
The Effect of a Web-Based Education Program and Educational Booklet Developed on Cervical Cancer on Women's Prevention Methods | 1.5 year
  To develop a web-based education program and an educational booklet on cervical cancer, and to assess the effectiveness of this program and booklet in improving women's knowledge, attitudes, and behaviors regarding cervical cancer prevention. The evaluation will be based on pre- and post-intervention surveys measuring changes in participants' understanding of cervical cancer, their attitudes toward screening and prevention, and their behaviors related to cervical cancer prevention practices.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sen, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Avcılar, Turkey (Türkiye)